CLINICAL TRIAL: NCT03632252
Title: Evaluating and Improving Assistive Robotic Devices Continuously and in Real-time
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never completed as planned.
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Deanna H Gates, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00139671; R03HD092639 (NIH)
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Powered ankle prosthesis (Experimental): We will use data from various sensors to optimize the amount of power provided by custom ankle ankle prosthesis. This is a single session study lasting about 4 hours.
  Interventions: Device: Powered ankle prosthesis

INTERVENTIONS:
Device: Powered ankle prosthesis — This device is a custom designed ankle prosthesis. Motors control force on the device through cables but are not worn by the person.

SUMMARY:
The goal of this research is to determine a quick, accurate and unobtrusive way to optimize the performance of powered assistive devices like ankle exoskeleton or prostheses.

DETAILED DESCRIPTION:
Lower limb assistive robotic devices, such as active prosthesis, orthoses, and exoskeletons have the potential to restore function for the millions of Americans who experience mobility challenges due to injury and disability. Since individuals with mobility challenges have an increased metabolic costs of transport, the benefit of such assistive devices is commonly assessed via the reduction in the metabolic work rate of the individual who is using the device. Currently, metabolic work rate can only be obtained in a laboratory environment, using breath-by-breath measurements of respiratory gas analysis. To obtain a single steady state data point of metabolic work rate, multiple minutes of data must be collected, since the signals are noisy and slow. In addition, the user has to wear a mask and bulky equipment. The investigators propose an improved way to obtain such estimates of metabolic work rate in real-time. In this project, the investigators will use various small sensors to optimize push-off timing for an active ankle prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Has a unilateral amputation
* Has used a prosthesis for at least 6 months

Exclusion Criteria:

* History of orthopedic or neurologic disorders to their intact limb
* History of cardiovascular disease
* Unable to walk for 30 minutes at a time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Minimum metabolic cost | 3 minutes
  The minimum oxygen consumption rate required for walking

CONTACTS AND LOCATIONS:
Overall Officials: Deanna H Gates, PhD, Principal Investigator — University of Michigan; C D Remy, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No